CLINICAL TRIAL: NCT00287820
Title: Independent Investigator Grant Study-Comparative Effects of Chronic Treatment With Olanzapine and Risperidone on Glucose and Lipid Metabolism
Brief Title: Comparative Effects of Chronic Treatment With Olanzapine and Risperidone on Glucose and Lipid Metabolism
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Nathan Kline Institute for Psychiatric Research (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Robert C. Smith MD, Manhatan Psychiatric Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FiD-MC-x226(7524)
Record Dates: First submitted 2006-02-06; First posted 2006-02-07 (Estimated); Last update posted 2011-07-25 (Estimated); Status verified 2007-12

CONDITIONS: Schizophrenia; Diabetes; Metabolic Syndrome; Hyperglycemia
Keywords: schizophrenia; diabetes; metabolic syndrome; hyperglycemia; glucose; insulin; lipids; IL-6; prolactin
MeSH Terms: conditions — Schizophrenia; Diabetes Mellitus; Metabolic Syndrome; Hyperglycemia; Insulin Resistance | interventions — Olanzapine; Risperidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): olanzapine
  Interventions: Drug: Olanzapine
- 2 (Active Comparator): risperidone
  Interventions: Drug: risperidone

INTERVENTIONS:
Drug: Olanzapine — olanzapine 5-40 mg/day
  Other Names: ayprexa
  Arms: 1
Drug: olanzapine — olanzapine 5-40 ,mg/day
  Other Names: zyprexa
  Arms: 1
Drug: risperidone — risperidone 1-12 mg/day
  Other Names: riperidal
  Arms: 2

SUMMARY:
The primary objective of the study is to assess whether chronic treatment with olanzapine over a five-month period produces a significant increase in abnormalities in glucose levels. The main secondary objective is to evaluate whether the increase in glucose levels and rate of glucose abnormalities differs between Olanzapine and Risperidone during this treatment period. Additional secondary objectives of the study are to investigate similar questions with respect to glycohemoglobin, triglycerides and other measures of glucose and lipid metabolism.

We hypothesize that Olanzapine will not be inferior to Risperidone in extent of increase in the primary outcome measure of serum glucose, and secondary measures of glycohemoglobin, insulin and lipids.

DETAILED DESCRIPTION:
In the on-going study in progress we use an extensive battery of assessments to investigate a)fasting levels of glucose and lipids at baseline and monthly during 5 months of treatment, b) glucose tolerance tests to investigate glucose and insulin abnormalities after a glucose load at baseline and during study treatment, and c)the effects of treatment with olanzapine and risperidone of post prandial glucose metabolism after a fatty meal (as detailed in the body of the proposal). Recent studies have shown that increased postprandial lipidemia is an important feature of many patients with type 2 diabetes and atherosclerosis. In addition to the biochemical measures, we will also assess clinical effects (PANSS and CGI ratings) and other side-effects (weight gain, appetite, somnolence, and EPS and TD). The specific plan calls for inpatients in a tertiary care hospital to be randomly assigned to olanzapine or risperidone, using a stratified random assignment procedure, and treated for five months with either olanzapine or risperidone. We estimate that we will have to enroll a sample of approximately 50-55 patients to obtain 46 acceptable complete cases(as specified in proposal below). On the basis of preliminary results from our prior and ongoing studies we predict no significant increase in glucose abnormalities from baseline during chronic treatment with olanzapine and no significant differences in development of glucose abnormalities in patients in patient treated with olanzapine and risperidone.

Additional measures being investigated include: comparison of olanzapine and risperidone in glucose and lipid responses to a fatty meal, ghrelin changes in response to a fatty mean, and CRP and IL-6, and thyroid and prolactin response to five months of treatment with the two drugs.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis
* Schizophrenia or schizoaffective psychosis
* 18-65 years of age

Exclusion Criteria:

* Currently being treated with oral antidiabetics or insulin

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2004-02; Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Serum glucose | during 5 months of treatment compared to baseline
Hb1AC | during 5 months of treatment compared to baseline
triglycerides | during 5 months of treatment compared to baseline
cholesterol | during 5 months of treatment compared to baseline
insulin | during 5 months of treatment compared to baseline
c-peptide | during 5 months of treatment compared to baseline

SECONDARY OUTCOMES:
ghrelin | during 5 months of treatment compared to baseline
CRP | during 5 months of treatment compared to baseline
Thyroid hormones | during 5 months of treatment compared to baseline
prolactin | during 5 months of treatment compared to baseline
Il-6 | during 5 months treatment compared to baseline
PANSS scores | during 5 months of treatment compared to baseline
CGI score | during 5 months of treatment compared to baseline
EPS scores | during 5 months of treatment compared to baseline
TD Scores | during 5 months of treatment compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Robert C Smith, MD PhD, Principal Investigator — NYU Medical School, Dept of Psychiatry and Manhattan Psychiatric Center
Locations (1):
- Manhattan Psychaitric Center, New York, New York, United States

REFERENCES:
- [Derived] Smith RC, Rachakonda S, Dwivedi S, Davis JM. Olanzapine and risperidone effects on appetite and ghrelin in chronic schizophrenic patients. Psychiatry Res. 2012 Oct 30;199(3):159-63. doi: 10.1016/j.psychres.2012.03.011. Epub 2012 Apr 3. PMID 22475524
- [Derived] Smith RC, Lindenmayer JP, Hu Q, Kelly E, Viviano TF, Cornwell J, Vaidhyanathaswamy S, Marcovina S, Davis JM. Effects of olanzapine and risperidone on lipid metabolism in chronic schizophrenic patients with long-term antipsychotic treatment: a randomized five month study. Schizophr Res. 2010 Jul;120(1-3):204-9. doi: 10.1016/j.schres.2010.04.001. Epub 2010 May 10. PMID 20457512
- [Derived] Smith RC, Lindenmayer JP, Davis JM, Kelly E, Viviano TF, Cornwell J, Hu Q, Khan A, Vaidhyanathaswamy S. Effects of olanzapine and risperidone on glucose metabolism and insulin sensitivity in chronic schizophrenic patients with long-term antipsychotic treatment: a randomized 5-month study. J Clin Psychiatry. 2009 Nov;70(11):1501-13. doi: 10.4088/JCP.08m04446yel. Epub 2009 Oct 6. PMID 19814947